CLINICAL TRIAL: NCT06417281
Title: A Phase III Clinical Trial of Photodynamic Diagnosis for Malignant Brain Glioma With 5-Aminolevulinic Acid
Brief Title: Photodynamic Diagnosis for Malignant Brain Glioma With 5-Aminolevulinic Acid（5-ALA）
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F0009-01
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-05

CONDITIONS: 5-aminolevulinic Acid; Malignant Glioma of Brain
MeSH Terms: interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5 Aminolevulinic Acid (Experimental): This is an single arm study.
  Interventions: Drug: 5 Aminolevulinic Acid

INTERVENTIONS:
Drug: 5 Aminolevulinic Acid — 3±1 hours before anesthesia, participants will take 5-ALA orally at a dosage of 20 mg/kg, followed by fluorescence-guided resection of malignant glioma.

SUMMARY:
This trial is an open-label, multicenter, phase III clinical study，conducted in patients with newly diagnosed or recurrent malignant high-grade (WHO grades 3~4) glioma, to evaluate the efficacy and safety of a single oral dose of 5-aminolevulinic acid (5-ALA) oral solution powder for fluorescence-guided tumor resection and photodynamic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient's written informed consent
* Age 18-75 years
* Radiological suspicion of a malignant glioma
* Indication for surgical tumour resection
* Karnofsky Performance Status (KPS) ≥ 70

Exclusion Criteria:

* Tumor located in the basal ganglia, thalamus, cerebellum, or brainstem
* Porphyria, hypersensitivity to porphyrins，history of cutaneous photosensitivity or photosensitive skin diseases；
* known hypersensitivity to the test drug ingredients
* Any other condition that, in the opinion of the investigator, makes participation in the trial inappropriate;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
positive predictive rate of tissue fluorescence per biopsy sample taken from fluorescent sites | within 48 hours after surgery
  The proportion of biopsy tissues diagnosed as malignant glioma cells positive by pathological examination among all tissues collected from both fluorescent and weakly fluorescent areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China